CLINICAL TRIAL: NCT03300817
Title: A Pilot Study of MUC1 Vaccine in Current and Former Smokers at High Risk for Lung Cancer
Brief Title: MUC1 Vaccine in Preventing Lung Cancer in Current and Former Smokers at High Risk for Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2017-01781; NCI-2017-01781 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N01-CN-2012-00042; MAY2016-08-01 (Other: Mayo Clinic in Rochester); MAY2016-08-01 (Other: DCP); N01CN00042 (NIH); P30CA015083 (NIH)
Record Dates: First submitted 2017-10-03; First posted 2017-10-04 (Actual); Results first posted 2023-04-19 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prevention (MUC1 peptide-Poly-ICLC vaccine) (Experimental): Patients receive MUC1 peptide-Poly-ICLC vaccine SC at weeks 0, 2, and 10.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: MUC1 Peptide-Poly-ICLC Vaccine

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: MUC1 Peptide-Poly-ICLC Vaccine — Given SC

SUMMARY:
This pilot phase I trial studies the side effects and how well MUC1 peptide-Poly-ICLC vaccine works in preventing lung cancer in current and former smokers at high risk for lung cancer. Vaccines made from peptides may help the body build an effective immune response to kill cells. MUC1 peptide-Poly-ICLC vaccine may stimulate the body's immune system and slow or stop the changes from normal to pre-cancer to cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Immunogenicity of the vaccine, assessed at week 12, based on the increase in IgG anti-MUC1 antibody titer over the pre-vaccination levels.

II. Safety, assessed throughout the trial and continued observation for 24 weeks.

SECONDARY OBJECTIVES:

I. To explore potential differences, if any, in the immunogenicity of the vaccine (as assessed at week 12 by the IgG anti-MUC1 antibody titer ratio) in current versus (vs.) former smokers.

II. To evaluate pre-vaccination levels of circulating myeloid derived suppressor cells (MDSC) and correlate with the ability to respond to the vaccine.

EXPLORATORY OBJECTIVES:

I. To explore immune response at week 24. II. To explore the relationship between chronic obstructive pulmonary disease (COPD) status at pre-registration and immune response in current versus former smokers.

III. To explore the impact of the MUC1 peptide-Poly-ICLC vaccine (MUC1/Poly-ICLC vaccine) on inflammation-related high sensitivity C-reactive protein (hsCRP) and interleukin-6 (IL-6) levels.

IV. To explore the impact of baseline levels of hsCRP and IL-6 on the ability to successfully vaccinate with MUC1/Poly-ICLC.

V. To establish a biospecimen repository archive: frozen peripheral blood live cells and plasma for future more detailed and comprehensive immunologic assays, including direct testing of anti-MUC1 T cell immunity.

OUTLINE:

Patients receive MUC1 peptide-Poly-ICLC vaccine subcutaneously (SC) at weeks 0, 2, and 10.

After completion of study treatment, patients may be followed up at week 28.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION INCLUSION CRITERIA
* Smoking history of >= 30 pack-years AND either current smoker (still smoking or quit < 1 year prior to pre-registration) OR former smoker (quit 1-15 years prior to pre-registration); Note: Pack years is determined by multiplying the number of packs smoked per day by the number of years smoked
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Computed tomography (CT) scan of the chest done =< 6 months prior to pre-registration showing either negative findings (no nodules) or solid or part-solid nodules < 6 mm in size (consistent with < 1% probability of malignancy, Lung-Reporting and Data Systems [RADs] version 1.0)
* Willingness to employ adequate contraception, if applicable; Note: women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* REGISTRATION INCLUSION CRITERIA
* Leukocytes (white blood cell [WBC]) >= 3,000/microliter
* Neutrophils (absolute neutrophil count [ANC]) >= 1,500/microliter
* Platelets >= 100,000/microliter
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) Note: Higher total bilirubin levels (=< 3 mg/dL) can be allowed if due to known benign liver condition, i.e. Gilbert's
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) =< 1.5 x institutional upper limit of normal (ULN)
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 x institutional upper limit of normal (ULN)
* Creatinine =< institutional upper limit of normal (ULN)

Exclusion Criteria:

* PRE-REGISTRATION EXCLUSION CRITERIA
* History of any malignancy; exceptions: non-melanoma skin cancer or carcinoma in situ (CIS) of the cervix
* Known hepatitis B or C
* Receiving any other investigational agents
* Any prior investigational immune therapy, such as for lung cancer prevention or treatment or for CIS of the cervix
* Use of oral or systemic steroids or other systemic anti-immune therapy =< 90 days prior to pre-registration; Note: Use of inhaled/nasal steroids and local steroid injections for pain control are not exclusionary
* Known human immunodeficiency virus (HIV)
* Known autoimmune disease
* Known non-alcoholic steatohepatitis (NASH) or non-alcoholic fatty liver disease (NAFLD)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MUC1/Poly-ICLC
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* REGISTRATION EXCLUSION CRITERIA
* Any positive antinuclear antibody (ANA) titer above 1:160, even in an asymptomatic individual. Note: Weakly positive ANA defined as ANA titers up to 1:160 maximum (=< 1:160) will be acceptable in an asymptomatic individual who is otherwise eligible for the study
* Pregnant or breast feeding; Note: Pregnant women are excluded from this study because the MUC1/Poly-ICLC vaccine may have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events (AEs) in nursing infants secondary to treatment of the mother with MUC1/Poly-ICLC vaccine, breastfeeding should be discontinued if the mother is treated with the vaccine

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2025-12-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Arjun Pennathur, Principal Investigator — Mayo Clinic in Rochester
Locations (2):
- United States (2):
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1 patient withdrew prior to beginning treatment and has been removed from all analyses
Period: Overall Study
Arm/Group | Prevention (MUC1 Peptide-Poly-ICLC Vaccine)
Started | 49
Completed | 45
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — Subject Found to be Ineligible | 2

BASELINE CHARACTERISTICS:
Arm/Group | Prevention (MUC1 Peptide-Poly-ICLC Vaccine)
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (4.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 48
  More than one race | 0
  Unknown or Not Reported | 0
Smoking Status [Count of Participants; unit: Participants]
  Current Smoker | 29
  Former Smoker | 20
Weight [Mean (Standard Deviation); unit: kg] | 83.1 (19.47)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Immunogenicity of the MUC1 Vaccine
Description: Will be evaluated by monitoring changes in IgG anti-MUC1 antibody titer ratio; defined as t12/t0, where t0 is the "initial titer" measured prior to vaccination, and t12 is the "final titer" drawn at 12 weeks. A titer ratio of >= 2 will be considered a positive response.
Time Frame: At week 12
Population: 4 patients are excluded from this analysis because they did not receive injections at weeks 2 and 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prevention (MUC1 Peptide-Poly-ICLC Vaccine)
Number analyzed (Participants) | 45
percentage of participants | 13.3 [5.1 to 26.8]

2. Primary Outcome: Count of Patients Experiencing 1 or More Grade 3+ Adverse Events at Least Possibly Related to Treatment
Description: Will be assessed according to National Cancer Institute Common Toxicity Criteria version 4.0. The maximum grade for each type of adverse event will be recorded for each participant and frequency tables will be reviewed to determine the overall patterns. In addition, the number and severity of adverse events will be tabulated and summarized across all grades.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prevention (MUC1 Peptide-Poly-ICLC Vaccine)
Number analyzed (Participants) | 49
Participants | 2

3. Secondary Outcome: Effect of Smoking Status on Vaccine Response
Description: To explore potential differences, if any, in the immunogenicity of the vaccine (as assessed at week 12 by the IgG anti-MUC1 antibody titer ratio) in current vs. former smokers.
Time Frame: 12 weeks
Measure: Number; unit: participants that responded to vaccine
Groups:
- Current Smoker: Patients that currently smoke
- Former Smoker: Patients that no longer smoke, but did in the past
Arm/Group | Current Smoker | Former Smoker
Number analyzed (Participants) | 27 | 18
participants that responded to vaccine | 4 | 2

4. Secondary Outcome: Pre-Vaccination Levels Versus Post-Vaccination Levels of Circulating Myeloid Derived Suppressor Cells (MDSC)
Description: Will correlate with the ability to respond to the vaccine. Will summarize the data using descriptive statistics and graphical methods (i.e. boxplots, scatter plots, etc.). For continuous MDSC data versus response data, will use t-tests or Wilcoxon Rank-Sum tests (for non-normal data).
Time Frame: 12 weeks
Population: Only patients with available data on levels of circulating myeloid derived suppressor cells at 12 weeks are included
Measure: Median (Full Range); unit: percent CD33
Groups:
- Non-Responder: Patients that did not experience a MUC1-specific IgG antibody titer that is ≥2 fold higher at 12 weeks compared to baseline
- Responder: Patients that experienced a MUC1-specific IgG antibody titer that is ≥2 fold higher at 12 weeks compared to baseline
Arm/Group | Non-Responder | Responder
Number analyzed (Participants) | 39 | 6
percent CD33 | 13.9 [1.4 to 37.9] | 9.4 [5.7 to 27.8]
Statistical Analysis 1: Comparison: Non-Responder vs Responder; Test type: Superiority; p = 0.6834, Wilcoxon Rank-Sum test

5. Other Pre Specified Outcome: Chronic Obstructive Pulmonary Disease (COPD) Status
Description: Will explore the relationship between COPD status at pre-registration and immune response in current versus former smokers. In individuals with COPD, the severity of airflow obstruction will be measured by the pulmonary function tests as per the GOLD classification.
Time Frame: Baseline to week 12
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Changes in Immunogenicity in Individuals With Chronic Obstructive Pulmonary Disease (COPD)
Description: Will explore whether or not changes in immunogenicity in individuals with COPD corresponds to different circulating MDSC levels.
Time Frame: Baseline up to week 12
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Impact of the MUC1/Poly-ICLC Vaccine on Inflammation-Related High Sensitivity C-Reactive Protein (hsCRP) and Interleukin-6 (IL-6)
Time Frame: Up to week 24
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Ability to Successfully Vaccinate With MUC1/Poly-ICLC Vaccine Depending on Baseline High Sensitivity C-Reactive Protein (hsCRP) and Interleukin-6 (IL-6) Levels
Time Frame: Up to week 24
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Prevention (MUC1 Peptide-Poly-ICLC Vaccine)
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 3/49
Other Adverse Events (participants affected / at risk) | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prevention (MUC1 Peptide-Poly-ICLC Vaccine) (N=49)
Hematuria (Renal and urinary disorders) | 1
Tooth infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prevention (MUC1 Peptide-Poly-ICLC Vaccine) (N=49)
Acidosis (Metabolism and nutrition disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Tooth infection (Infections and infestations) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Urinary tract infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 4
Transient ischemic attacks (Nervous system disorders) | 1
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 3
Skin infection (Infections and infestations) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Serum amylase increased (Investigations) | 5
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pain (General disorders) | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Lipase increased (Investigations) | 5
Leukocytosis (Blood and lymphatic system disorders) | 1
Investigations - Other, specify (Investigations) | 4
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1
Injection site reaction (General disorders) | 37
Infections and infestations - Other, specify (Infections and infestations) | 2
Immune system disorders - Other, specify (Immune system disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Headache (Nervous system disorders) | 4
Hematuria (Renal and urinary disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 5
Gastritis (Gastrointestinal disorders) | 1
Forced expiratory volume decreased (Investigations) | 1
Flu like symptoms (Gastrointestinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Eye disorders - Other, specify (Eye disorders) | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Edema face (General disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 2
Creatinine increased (Investigations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Allergic reaction (Immune system disorders) | 1
Alkaline phosphatase increased (Investigations) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/17/NCT03300817/Prot_SAP_ICF_001.pdf